CLINICAL TRIAL: NCT03245450
Title: A Phase 1/2 Single-arm Study Evaluating the Safety and Efficacy of Eribulin Mesilate in Combination With Irinotecan in Children With Refractory or Recurrent Solid Tumors
Brief Title: Study Evaluating the Safety and Efficacy of Eribulin Mesilate in Combination With Irinotecan Hydrochloride in Children With Refractory or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-213; 2016-003352-67 (EudraCT Number)
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2021-06

CONDITIONS: Refractory or Recurrent Solid Tumors; Rhabdomyosarcoma; Non-Rhabdomyosarcoma Soft Tissue Sarcoma; Ewing Sarcoma
Keywords: eribulin mesilate; irinotecan; combination therapy; children
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma; Sarcoma, Ewing | interventions — eribulin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eribulin mesilate plus irinotecan hydrochloride (Experimental): In Schedules A and B, eribulin mesilate at the dose of 1.4 milligrams per meters squared (mg/m^2) will be administered as an intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle. In Schedule A, irinotecan hydrochloride at the doses of 20 mg/m^2 or 40 mg/m^2 will be administered as an IV infusion on Days 1 to 5 of a 21-day cycle. In Schedule B, irinotecan hydrochloride at the doses of 100 mg/m^2 or 125 mg/m^2 will be administered as an IV infusion on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Eribulin mesilate; Drug: Irinotecan hydrochloride

INTERVENTIONS:
Drug: Eribulin mesilate — IV infusion
  Other Names: E7389
Drug: Irinotecan hydrochloride — IV infusion
  Other Names: (S)-4,11-diethyl-39 3,4,12,14-tetrahydro-4-hydroxy-3,14-dioxo-1H-pyrano[3',4':6,7]-indolizino[1,2-b]quinolin-9-4-yl-[1,4'-bipiperidine]-1'-carboxylate, monohydrochloride, trihydrate

SUMMARY:
The Phase 1 part of the study is conducted to determine the maximum tolerated dose (MTD) and Recommended Phase 2 Dose (RP2D) of eribulin mesilate in combination with irinotecan hydrochloride in pediatric participants with relapsed/refractory solid tumors (excluding central nervous system [CNS] tumors).

The Phase 2 part of the study is conducted to assess the objective response rate (ORR) and duration of response (DOR) of eribulin mesilate in combination with irinotecan hydrochloride in pediatric participants with relapsed/refractory rhabdomyosarcoma (RMS), non-rhabdomyosarcoma soft tissue sarcoma (NRSTS) and ewing sarcoma (EWS).

ELIGIBILITY:
Participants must be

* >=12 months to less than or equal to (<=) 25 years old at the time of consent [no more than 25 percent (%) of participants between the ages of 18 and 25 years will be enrolled in this study].
* In Phase 1, >6 months and <12 months at the time of consent (Schedule A only) participants will be enrolled one dose level behind the >=12 months participant in order to maximize safety for infant participants. In Phase 2, participants aged >6 months and <12 months at the time of consent will be enrolled to Schedule A with a modified dose of eribulin with the irinotecan dose maintained in order to maximize safety for infant participants.

Inclusion Criteria:

* Phase 1: Participants must be diagnosed with histologically confirmed solid tumors (excluding CNS tumors), which is relapsed or refractory, and for which there are no currently available therapies.
* Phase 2: Participants must be diagnosed with histologically confirmed RMS, NRSTS or EWS which is relapsed or refractory having received at least 1 prior therapy, including primary treatment.
* Phase 1: Participants must have either measurable or evaluable disease as per RECIST 1.1.
* Phase 2: Participants must have measurable disease as per RECIST 1.1.
* Participant's current disease state must be one for which there is no known curative therapy.
* Participant's performance score must be >=50% Karnofsky (for participants >16 years of age) or Lansky (for participants <=16 years of age).Participants who are unable to walk because of paralysis and/or previous surgeries, but who are in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participants must have fully recovered from the acute toxic effects of all prior anticancer treatments prior to study drug administration:

  * Must not have received myelosuppressive chemotherapy within 21 days prior to study drug administration (42 days if prior nitrosourea).
  * Must not have received a long-acting growth factor (example, Neulasta) within 14 days or a short-acting growth factor within 7 days.
  * Must not have received an antineoplastic targeted therapy within 14 days.
  * Must not have received immunotherapy, example, tumor vaccines, within 42 days.
  * Must not have received monoclonal antibodies within at least 3 half-lives of the antibody after its last dose.
  * Must not have received radiotherapy (XRT) within 14 days prior to study drug administration (small field) or 42 days for craniospinal XRT, or if >=50% radiation of pelvis.
  * At least 84 days must have elapsed after stem cell infusion prior to study drug administration
  * No evidence of active graft-versus-host disease (GVHD) and at least 100 days must have elapsed after allogeneic bone marrow transplant or stem cell infusion prior to study drug administration
* Participants must have adequate bone marrow function, defined as:

  * Peripheral absolute neutrophil count (ANC) >=1.0*10^9/liter (L).
  * Platelet count >=100*10^9/L (not receiving platelet transfusions within a 7-day period prior to study drug administration).
  * Hemoglobin (Hb) at least 8.0 grams per deciliter (g/dL) at baseline (blood transfusions are allowed during the screening period to correct Hb values <8.0 g/dL).
* Participants must have adequate renal function, defined as:

  * A serum creatinine based on age/gender, derived from the Schwartz formula for estimating glomerular filtration rate (GFR), per protocol-specified criteria.
  * Serum creatinine clearance or GFR >=50 milliliters/minute/1.73 m^2, based on a 12 or 24 hours (h) urine creatinine collection.
* Participants must have adequate liver function, defined as:

  * Bilirubin (sum of conjugated + unconjugated) <=1.5 times the upper limit of normal (ULN) for age.
  * Alkaline phosphatase, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3*ULN (in the case of liver metastases <=5*ULN), unless there are bone metastases, in which case liver-specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
  * Serum albumin >=2 g/dL.
* All participants and/or their parents or guardians must sign a written informed consent.
* Participants must be willing to comply with all aspects of the protocol.

Exclusion Criteria:

* Females who are breastfeeding or pregnant at Screening or Baseline. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 h before the first dose of study drug.
* Females of childbearing potential who:

  * Do not agree to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation, that is:
  * Total abstinence (if it is their preferred and usual lifestyle)
  * An intrauterine device (IUD) or intrauterine system (IUS)
  * A contraceptive implant
  * An oral contraceptive OR
  * Do not have a vasectomized partner with confirmed azoospermia.
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period or for 3 months after study drug discontinuation). No sperm donation is allowed during the study period or for 3 months after study drug discontinuation.
* Concomitant Medications:

  * Participants receiving corticosteroids who have not been on a stable dose for at least 7 days prior to study drug administration.
  * Participants who are currently receiving other anticancer agents.
  * Participants who are receiving cyclosporine, tacrolimus or other agents to prevent GVHD post bone marrow transplant.
  * Participants who are receiving strong cytochrome P450 3A4 (CYP3A4) inhibitors and inducers including traditional herbal medicinal products (example, St. John's Wort).
* Phase 1: Received prior therapy with eribulin mesilate within 6 months prior to study drug administration.
* Phase 2: Received prior therapies with eribulin mesilate or irinotecan hydrochloride (for prior irinotecan hydrochloride, participants can be included if there was no tumor progression during irinotecan therapy).
* Any other malignancy that required treatment (except non-melanoma skin cancer, or histologically confirmed complete excision of carcinoma in situ), within 2 years prior to study drug administration.
* Has hypersensitivity to either study drug or any of the excipients.
* Has a known prior history of viral hepatitis (B or C) as demonstrated by positive serology (presence of antigens) or have an uncontrolled infection requiring treatment
* Has >Grade 1 peripheral sensory neuropathy or >Grade 1 peripheral motor neuropathy graded according to the Modified ("Balis") Pediatric Scale of Peripheral Neuropathies.
* Has cardiac pathology, defined as:

  * Participants with known congestive heart failure, symptomatic or Left ventricular (LV) ejection fraction <50% or shortening fraction <27% and participants with congenital long QT syndrome, bradyarrhythmias, or QT interval (QTc)>480 milliseconds on at least 2 separate electrocardiograms (ECGs).
* Has CNS disease: Participants with brain or subdural metastases are not eligible unless the metastases are asymptomatic and do not require treatment or have been adequately treated by local therapy and have discontinued the use of corticosteroids for this indication for at least 28 days prior to study drug administration. Participants must be clinically stable. It is not the intention of this protocol to treat participants with active brain metastases.

Note: Screening CNS imaging for participants with a known history of CNS disease is required.

* Have had or are planning to have the following invasive procedures:

  * Major surgical procedure or significant traumatic injury within 28 days prior to study drug administration.
  * Laparoscopic procedure or open biopsy within 7 days prior to study drug administration
  * Central line placement or subcutaneous port placement is not considered major surgery.
  * Core biopsy, including bone marrow biopsy within 2 days prior to study drug administration.
  * Fine needle aspirate within 3 days prior to study drug administration.
* Participants with known human immunodeficiency virus (HIV); due to lack of available safety data for eribulin therapy in HIV infected participants.
* Has any serious concomitant illness that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments (including active or severe chronic inflammatory bowel disease or bowel obstruction).
* Has received a live-virus vaccination within 30 days of planned start of study therapy. Seasonal flu vaccines that do not contain live virus are permitted.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- France (3):
  - Hopitaux de La Timone, Marseille, Bouches-du-Rhône
  - Centre Oscar Lambret, Lille, Nord
  - Centre Léon Berard, Lyon, Rhône
- Germany (6):
  - Eisai Trial Site 4, Freiburg im Breisgau, Baden-Wurttemberg
  - Eisai Trial Site 2, Frankfurt am Main, Hesse
  - Eisai Trial Site 5, Göttingen, Lower Saxony
  - Eisai Trial Site 1, Aachen, North Rhine-Westphalia
  - Eisai Trial Site 3, Berlin
  - Eisai Trial Site 6, Essen
- Greece (2):
  - Aghia Sophia' Children's General Hospital of Athens, Athens, Attica
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
- Italy (8):
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Istituto G Gaslini Ospedale Pediatrico IRCCS, Genoa, Liguria
  - Ospedale Infantile Regina Margherita, Turin, Piedmont
  - Azienda Ospedaliera A Meyer, Florence, Tuscany
  - Azienda Ospedaliera Di Padova, Padua, Veneto
  - Istituto Nazionale Dei Tumori, Milan
- Poland (2):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Masovian Voivodeship
- Spain (6):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Kinderspital Zürich - Eleonorenstiftung, Zurich, Switzerland
- United Kingdom (11):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Southampton General Hospital, Southampton, Hampshire
  - Alder Hey Childrens Hospital, Liverpool, Merseyside
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital - Surrey, Sutton, Surrey
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - The Leeds Teaching Hospitals Charitable Foundation - Leeds Childrens Hospital (LCH), Leeds, Yorkshire
  - University College London, London
  - Royal Manchester Childrens Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester
  - Royal Victoria Infirmary, Newcastle

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 22 investigative sites in France, Germany, Greece, Italy, Poland, Spain and United Kingdom from 05 March 2018 to 17 May 2021.
Pre-assignment Details: A total of 46 participants were screened, out of which 13 participants were treated in the Phase 1 and 27 participants were treated in Phase 2 (9 participants each in the relapsed/refractory rhabdomyosarcoma [RMS], non-rhabdomyosarcoma soft tissue sarcoma [NRSTS], and Ewing sarcoma [EWS] cohorts).
Groups:
- Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2: Participants received eribulin mesilate 1.4 mg/m^2 (milligram per square meter) intravenous infusion on Days 1 and 8 and irinotecan hydrochloride 20 mg/m^2, intravenous infusion on Days 1 to 5 in every 21 days treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
- Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2: Participants received eribulin mesilate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and irinotecan hydrochloride 40 mg/m^2, intravenous infusion on Days 1 to 5 in every 21 days treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
- Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2: Participants received eribulin mesilate 1.4 mg/m^2 and irinotecan hydrochloride 100 mg/m^2 intravenous infusion on Days 1 and 8 in every 21 days treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
- Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2: Participants received eribulin mesilate 1.4 mg/m^2 and irinotecan hydrochloride 125 mg/m^2 intravenous infusion on Days 1 and 8 in every 21 days treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
- Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2: Participants with RMS received eribulin mesilate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and irinotecan hydrochloride 40 mg/m^2, intravenous infusion on Days 1 to 5 in every 21 days treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
- Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2: Participants with NRSTS received eribulin mesilate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and irinotecan hydrochloride 40 mg/m^2, intravenous infusion on Days 1 to 5 in every 21 days treatment cycle until disease progression, development of unacceptable toxicity or withdrawal of consent.
- Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2: Participants with EWS received eribulin mesilate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and Irinotecan hydrochloride 40 mg/m^2, intravenous infusion on Days 1 to 5 in every 21 days treatment cycle until disease progression, development of unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
Started | 3 | 4 | 3 | 3 | 9 | 9 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 3 | 9 | 9 | 9
Not completed — Radiological disease progression | 3 | 3 | 2 | 2 | 7 | 6 | 6
Not completed — Clinical disease progression | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of either study drug.
Groups:
- Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2: Participants received eribulin mesilate 1.4 mg/m^2 intravenous infusion on Days 1 and 8 and irinotecan hydrochloride 20 mg/m^2, intravenous infusion on Days 1 to 5 in every 21 days treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 9 | 9 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per the planned analysis, baseline data for participants in Phase 1 and Phase 2 were not combined, therefore Mean and Standard Deviation are presented separately for Phase 1 and Phase 2 participants.
  years
    Phase 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 0 | 0 | 0 | 13
    Phase 1 | 10.94 (6.583) | 7.33 (2.540) | 13.97 (4.231) | 8.06 (4.997) |  |  |  | 9.87 (4.842)
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9 | 9 | 27
    Phase 2 |  |  |  |  | 11.05 (3.845) | 12.71 (4.348) | 11.59 (3.753) | 11.78 (3.899)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 1 | 4 | 1 | 2 | 5 | 3 | 4 | 20
  Adolescents (12-17 years) | 2 | 0 | 2 | 1 | 4 | 6 | 5 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 5 | 2 | 5 | 19
  Male | 1 | 3 | 1 | 1 | 4 | 7 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 9 | 8 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 4 | 2 | 3 | 5 | 8 | 8 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D) of Eribulin Mesilate in Combination With Irinotecan Hydrochloride
Description: The RP2D was evaluated based on a review of the outcomes of safety (including dose limiting toxicities [DLTs]), tumor assessments, and pharmacokinetic (PK) in Phase 1 by investigators and the study team.
Time Frame: First dose of study drug up to Cycle 1 (Cycle length=21 days)
Population: The Dose Evaluable Set (DES) for Phase 1 included all the participants who completed Cycle 1 treatment and were evaluated for DLTs and those who discontinued treatment during Cycle 1 due to DLTs.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: All Participants: All participants received eribulin mesilate 1.4 mg/m^2 intravenous infusion on Days 1 and 8 and irinotecan hydrochloride 20 mg/m^2 or 40 mg/m^2 intravenous infusion on Days 1 to 5 (schedule A) and irinotecan hydrochloride 100 mg/m^2 or 125 mg/m^2 intravenous infusion on Days 1 and 8 (schedule B) in 21-day treatment cycle until disease progression, development of intolerable toxicity or withdrawal of consent.
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 12
mg/m^2
  Eribulin Mesilate | 1.4
  Irinotecan Hydrochloride | 40

2. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving best overall response (BOR) of confirmed partial response (PR) or complete response (CR) determined by investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have a reduction in their short axis less than (<) 10 millimeter (mm). PR was at least a 30 percent (%) decrease in the sum of diameter (SOD) of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or up to approximately 2 years 4 months
Population: Full analysis set included all participants who received at least 1 dose of either study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
Number analyzed (Participants) | 9 | 9 | 9
percentage of participants | 11.1 (0.6) [0.6 to 42.9] | 11.1 (0.6) [0.6 to 42.9] | 11.1 (0.6) [0.6 to 42.9]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an AE that emerged during treatment, having been absent at pretreatment, or reemerged during treatment, having been present at pre-treatment (baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous. AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: From first dose of study drug up to approximately 2 years 4 months
Population: Safety analysis set included all participants who received at least 1 dose of either study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 9 | 9
Participants | 3 | 4 | 3 | 3 | 9 | 9 | 9

4. Secondary Outcome: Number of Participants With Serious Adverse Event (SAE)
Description: SAE was defined as any untoward medical occurrence at any dose if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: Up to approximately 2 years and 4 months
Population: Safety analysis set included all participants who received at least 1 dose of either study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 9 | 9
Participants | 1 | 3 | 0 | 1 | 5 | 4 | 3

5. Secondary Outcome: Phase 1, Cmax: Maximum Observed Plasma Concentration of Eribulin, Irinotecan and Its Active Metabolite SN-38
Time Frame: For eribulin, Cycle 1 Day 1: 0-120 hours post-eribulin infusion; For irinotecan and its metabolite, Cycle 1 Day 1: 0-24 hours post-irinotecan infusion (cycle length=21 days)
Population: PK analysis set included participants who had documented dosing history and at least one post-dosing quantifiable drug concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 4 | 3 | 3
nanogram/milliliter (ng/mL)
  Eribulin | 369.3 (58.0) [lower limit 58.0] | 179.4 (136.1) [lower limit 136.1] | 348.7 (25.0) [lower limit 25.0] | 323.3 (20.6) [lower limit 20.6]
  Irinotecan | 538.8 (165.9) [lower limit 165.9] | 399.5 (19.1) [lower limit 19.1] | 1168.1 (39.8) [lower limit 39.8] | 1555.4 (39.5) [lower limit 39.5]
  Active Metabolite SN-38 | 6.518 (9.4) [lower limit 9.4] | 17.170 (39.7) [lower limit 39.7] | 25.409 (51.6) [lower limit 51.6] | 18.614 (74.3) [lower limit 74.3]

6. Secondary Outcome: Phase 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of Eribulin, Irinotecan and Its Active Metabolite SN-38
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 4 | 3 | 3
hours
  Eribulin | 0.080 (0.03) [0.03 to 0.22] | 0.135 (0.03) [0.03 to 1] | 0.080 (0) [0 to 0.12] | 0.050 (0.01) [0.01 to 0.12]
  Irinotecan | 0.250 (0.07) [0.07 to 0.42] | 0.305 (0) [0 to 24] | 0.300 (0.03) [0.03 to 0.33] | 0.170 (0.13) [0.13 to 0.25]
  Active Metabolite SN-38 | 0.420 (0.25) [0.25 to 1.03] | 0.305 (0) [0 to 24] | 0.330 (0.3) [0.3 to 0.53] | 0.250 (0.13) [0.13 to 0.55]

7. Secondary Outcome: Phase 1, T1/2: Half-life of Eribulin, Irinotecan and Its Active Metabolite SN-38
Description: Half-life for irinotecan and metabolite SN-38 could not be estimated for phase 1:schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 20 mg/m^2 and phase 1: schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 40 mg/m^2 arm as the slope of the terminal phase of the concentration-time profiles could not be determined.
Time Frame: as for outcome 5
Population: PK analysis set included participants who had documented dosing history and at least one post-dosing quantifiable drug concentration. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure and 'n' (number analyzed) included all participants who were evaluable for each category.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 2
hours
  Eribulin | 27.50 [26.5 to 27.7] | 34.70 [32.9 to 40.4] | 30.00 [23.4 to 43.3] | 25.30 [22.1 to 28.5]
  Irinotecan: number analyzed (Participants) | 0 | 0 | 3 | 2
  Irinotecan |  |  | 5.140 [5.1 to 9.61] | 4.430 [3.95 to 5.08]
  Metabolite SN-38: number analyzed (Participants) | 0 | 0 | 3 | 2
  Metabolite SN-38 |  |  | 12.000 [9.9 to 13.9] | 10.390 [9.68 to 11.1]

8. Secondary Outcome: Phase 1, Total Clearance (CL) of Eribulin and Irinotecan
Description: CL for irinotecan could not be estimated for phase 1:schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 20 mg/m^2 and phase 1: schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 40 mg/m^2 arm because it was not possible to calculate half-life as the slope of the terminal phase of the concentration-time profiles could not be determined.
Time Frame: For eribulin, Cycle 1 Day 1: 0-120 hours post-eribulin infusion; For irinotecan, Cycle 1 Day 1: 0-24 hours post-irinotecan infusion (cycle length=21 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 2
liter per hour (L/h)
  Eribulin | 3.1781 (43.9) | 2.4581 (8.0) | 2.9060 (32.8) | 1.7521 (136.6)
  Irinotecan: number analyzed (Participants) | 0 | 0 | 3 | 2
  Irinotecan |  |  | 27.27 (23.2) | 30.30 (60.7)

9. Secondary Outcome: Phase 1, Volume of Distribution (Vz) of Eribulin and Irinotecan
Description: Vz for irinotecan could not be estimated for phase 1: schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 20 mg/m^2 and phase 1: schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 40 mg/m^2 arm because it was not possible to calculate half-life as the slope of the terminal phase of the concentration-time profiles could not be determined.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 2
liter
  Eribulin | 124.70 (41.5) | 126.96 (18.1) | 130.78 (35.9) | 63.35 (101.8)
  Irinotecan: number analyzed (Participants) | 0 | 0 | 3 | 2
  Irinotecan |  |  | 248.5 (16.1) | 195.1 (69.0)

10. Secondary Outcome: Phase 1, AUC(0-t): Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration of Eribulin, Irinotecan and Its Active Metabolite SN-38
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 4 | 3 | 3
hour*nanogram per milliliter (h*ng/mL)
  Eribulin | 422.5 (40.0) [lower limit 40.0] | 403.7 (32.1) [lower limit 32.1] | 616.9 (66.1) [lower limit 66.1] | 603.5 (87.3) [lower limit 87.3]
  Irinotecan | 1812.6 (13.5) [lower limit 13.5] | 3686.1 (36.4) [lower limit 36.4] | 4693.9 (66.1) [lower limit 66.1] | 3633.7 (38.9) [lower limit 38.9]
  Metabolite SN-38 | 68.00 (19.7) [lower limit 19.7] | 145.04 (11.6) [lower limit 11.6] | 138.22 (42.2) [lower limit 42.2] | 65.47 (153.2) [lower limit 153.2]

11. Secondary Outcome: Phase 1, AUC(0-inf): Area Under the Concentration-time Curve From Zero (Pre-dose) Extrapolated to Infinite Time of Eribulin, Irinotecan and Its Active Metabolite SN-38
Description: AUC(0-inf) for irinotecan and metabolite SN-38 could not be estimated for phase 1: schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 20 mg/m^2 and phase 1: schedule A, eribulin mesilate 1.4 mg/m^2 + irinotecan 40 mg/m^2 arm because it was not possible to calculate half-life as the slope of the terminal phase of the concentration-time profiles could not be determined.
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 2
h*ng/mL
  Eribulin | 438.1 (39.0) | 506.0 (16.6) | 666.9 (69.0) | 576.9 (133.6)
  Irinotecan: number analyzed (Participants) | 0 | 0 | 3 | 2
  Irinotecan |  |  | 5036.1 (70.9) | 3698.5 (39.2)
  Metabolite SN-38: number analyzed (Participants) | 0 | 0 | 3 | 2
  Metabolite SN-38 |  |  | 169.0 (51.4) | 149.4 (4.3)

12. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the date of disease progression (PD). PFS was assessed based on the investigators' assessments utilizing RECIST 1.1. PD was defined as at least 20% increase or 5 mm increase in the sum of diameters of target lesions recorded since the treatment started or the appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan-Meier method.
Time Frame: From the date of first dose to the date of first documentation of PD, or date of death, whichever occurred first up to approximately 2 years 4 months
Population: Full analysis set included all participants who received at least 1 dose of either study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
Number analyzed (Participants) | 9 | 9 | 9
months | 2.69 (1.28) [1.28 to 8.87] | 1.35 (1.15) [1.15 to 2.79] | 6.70 (1.38) [1.38 to 8.84]

13. Secondary Outcome: Phase 2: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with BOR of CR, PR, or durable stable disease (SD) based on RECIST 1.1 (durable SD was defined as SD with duration of greater than [>] 11 weeks). CR was defined as disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have a reduction in their short axis <10 mm. PR was defined as at least 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 12
Population: Full analysis set included all participants who received at least 1 dose of either study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
Number analyzed (Participants) | 5 | 3 | 5
percentage of participants | 55.6 (25.1) [25.1 to 83.1] | 33.3 (9.8) [9.8 to 65.5] | 55.6 (25.1) [25.1 to 83.1]

14. Secondary Outcome: Model Predicted Apparent Total Body Clearance (CL) of Eribulin
Description: Per the planned PK analysis, PK samples were collected and analyzed using a population PK approach to estimate PK parameters. Eribulin plasma concentration data from this study were pooled from studies (NCT00069264, NCT00069277, NCT00326950, NCT00706095, NCT01000376, NCT01106248, NCT02171260, NCT00413192, NCT01458249, NCT03441360 and NCT01327885), and a population PK model was applied to the pooled dataset. The data presented are the CL parameter estimates, with Measure Type "Number" defining the eribulin PK model. They are population PK model predictions and have been estimated using non-linear mixed effects model.
Time Frame: Cycle 1 Day 1: 0.5-120 hours after eribulin infusion; Cycle 1 Day 8: pre-dose and at the end of the eribulin infusion (cycle length=21 days)
Population: PK analysis set included all participants who had documented dosing history had at least one postdosing quantifiable drug concentration. Analysis population for this outcome measure included participants from current study E7389-G000-213 and from studies (NCT00069264,NCT00069277,NCT00326950,NCT00706095,NCT01000376,NCT01106248,NCT02171260, NCT00413192,NCT01458249,NCT03441360,NCT01327885)."Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: L/hr
Groups:
- Eribulin Mesilate - All Participants: All participants who received eribulin mesilate intravenous infusion over the dose range 0.25 to 4.0 mg/m^2 in current study (E7389-G000-213) and studies (NCT00069264, NCT00069277, NCT00326950, NCT00706095, NCT01000376, NCT01106248, NCT02171260, NCT00413192, NCT01458249, NCT03441360 and NCT01327885).
Arm/Group | Eribulin Mesilate - All Participants
Number analyzed (Participants) | 561
L/hr | 2.89 [2.75 to 3.03]

15. Secondary Outcome: Volume of Distribution Estimates From the Population PK Model for Eribulin
Description: Per the planned PK analysis, PK samples were collected and analyzed using a population PK approach to estimate PK parameters. Eribulin plasma concentration data from this study were pooled from studies (NCT00069264, NCT00069277, NCT00326950, NCT00706095, NCT01000376, NCT01106248, NCT02171260, NCT00413192, NCT01458249, NCT03441360 and NCT01327885), and a population PK model was applied to the pooled dataset. Data presented are the volume of distribution of the central compartment (V1), volume of distribution of the first peripheral compartment (V2), and volume of distribution of the second peripheral compartment (V3) parameter estimates with Measure Type "Number" defining the eribulin PK model. They are population PK model predictions and have been estimated using non-linear mixed effects model.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: liter
Groups:
- Eribulin Mesilate - All Participants: All participants who received eribulin mesilate intravenous infusion over the dose range 0.25 to 4.0 mg/m^2 in current study (E7389-G000-213) and in studies (NCT00069264, NCT00069277, NCT00326950, NCT00706095, NCT01000376, NCT01106248, NCT02171260, NCT00413192, NCT01458249, NCT03441360 and NCT01327885).
Arm/Group | Eribulin Mesilate - All Participants
Number analyzed (Participants) | 561
liter
  V1 | 4.08 [3.87 to 4.29]
  V2 | 2.03 [1.79 to 2.27]
  V3 | 106 [101 to 111]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 2 year 4 months
Arm/Group | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/4 | 1/3 | 1/3 | 4/9 | 3/9 | 3/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/4 | 0/3 | 1/3 | 5/9 | 4/9 | 3/9
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 3/3 | 9/9 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 (N=3) | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=4) | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 (N=3) | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 (N=3) | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=9) | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=9) | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=9)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 20 mg/m^2 (N=3) | Phase 1: Schedule A, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=4) | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 100 mg/m^2 (N=3) | Phase 1: Schedule B, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 125 mg/m^2 (N=3) | Phase 2: RMS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=9) | Phase 2: NRSTS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=9) | Phase 2: EWS Cohort, Eribulin Mesilate 1.4 mg/m^2 + Irinotecan 40 mg/m^2 (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (14) | 1 (6) | 1 (1) | 3 (9) | 4 (8) | 5 (29)
Leukopenia (Blood and lymphatic system disorders) | 1 (4) | 1 (14) | 2 (15) | 1 (12) | 0 (0) | 1 (1) | 3 (32)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (39) | 2 (8) | 3 (18) | 1 (12) | 3 (15) | 2 (10) | 4 (52)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (17)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 2 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (12) | 0 (0) | 0 (0) | 4 (24) | 5 (11) | 5 (9)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 6 (8) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (10) | 1 (3) | 6 (8) | 2 (2) | 1 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 5 (8)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (10) | 1 (2) | 2 (9)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (5)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (8) | 0 (0) | 2 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (8) | 0 (0) | 2 (7) | 6 (21) | 3 (22) | 5 (46)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 3 (7) | 0 (0) | 1 (1) | 1 (20) | 1 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (4)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (3) | 2 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0)
Metamyelocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 2 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Refeeding syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 2 (5)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Negative thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tearfulness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukonychia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT03245450/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT03245450/SAP_001.pdf